CLINICAL TRIAL: NCT03643224
Title: A Prospective Clinical Evaluation of the DiamondTemp™ System for the Treatment of Persistent Atrial Fibrillation
Brief Title: DiamondTemp™ System for the Treatment of Persistent Atrial Fibrillation
Acronym: Diamond-AFII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP01071
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Persistent Atrial Fibrillation; Atrial Fibrillation
Keywords: ablation; electrophysiology; atrial fibrillation; catheter; persistent
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Experimental (Experimental): Radiofrequency Ablation. Catheter ablation to treat persistent atrial fibrillation using temperature-controlled ablation catheter
  Interventions: Device: Radiofrequency Ablation

INTERVENTIONS:
Device: Radiofrequency Ablation — A procedure will be performed using a radiofrequency ablation catheter.

SUMMARY:
The purpose of the Diamond-AF II study is to establish the safety and effectiveness of the DiamondTemp Ablation System for the treatment of drug refractory, symptomatic persistent atrial fibrillation in patients.

DETAILED DESCRIPTION:
The DIAMOND-AF II Study is a prospective, non-randomized (single-group assignment) trial being performed at multiple centers in the United States, Canada and Europe to evaluate the safety and effectiveness of the DiamondTemp Ablation System for the treatment of patients with persistent atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Above eighteen (18) years of age or of legal age to give informed consent specific to state and national law.
2. Subjects with a history of documented symptomatic, persistent Atrial Fibrillation with 1) a physician's note documenting a continuous AF episode lasting longer than 7 days but less than 12 months AND 2) two electrocardiograms from any form of rhythm monitoring showing continuous AF taken at least 7 days apart OR a 24-hour Holter within 180 days of the ablation procedure showing continuous AF.
3. Refractory, intolerant or contraindicated to at least one Class I or III anti-arrhythmic (AAD) drug.
4. Suitable candidate for intra-cardiac mapping and ablation of arrhythmia.
5. Subject agrees to comply with study procedures and be available (geographically stable) for follow-up visits for at least 12 months after enrollment.
6. Subject is willing and able to provide written consent.

Exclusion Criteria:

At time of enrollment and/or prior to procedure:

1. Continuous AF >12 months (long-standing persistent AF)
2. Paroxysmal AF with longest episode <7 days
3. AF secondary to electrolyte imbalance, thyroid disease or reversible or non-cardiac cause
4. Rheumatic heart disease
5. Severe mitral regurgitation
6. Hypertrophic cardiomyopathy
7. LA diameter >5.5 cm
8. Left ventricular ejection fraction (LVEF) <40%
9. Currently NYHA Class III or IV or exhibits uncontrolled heart failure
10. Body Mass Index (BMI) >42 kg/m2.
11. LA ablation, septal closure device or mitral valve surgical procedure at any time prior to enrollment
12. Presence of intramural thrombus, tumor or abnormality that precludes vascular access, catheter introduction or manipulation
13. Coagulopathy, bleeding diathesis or suspected procoagulant state
14. Sepsis, active systemic infection or fever (>100.5 oF / 38 oC) within a week prior to the ablation procedure
15. Significant restrictive or obstructive pulmonary disease or chronic respiratory condition
16. Renal failure requiring dialysis or renal compromise that in the investigator's judgement would increase risk to the subject or deem the subject inappropriate to participate in the study.
17. Known allergies or intolerance to anticoagulant and antiplatelet therapies to be used in conjunction with the study or contrast sensitivity that cannot be adequately pre-treated prior to the ablation procedure.
18. Positive pregnancy test results for female subjects of childbearing potential or breast feeding.
19. Enrollment in a concurrent clinical study that in the judgement of the investigator would impact study outcomes.
20. Acute or chronic medical condition that in the judgment of the investigator would increase risk to the subject or deem the subject inappropriate to participate in the study.
21. Life expectancy <12 months based on medical history or the medical judgement of the investigator.

    Within 1 month of enrollment or just prior to procedure:
22. Documented LA thrombus upon imaging
23. Creatinine >2.5mg/dl or creatinine clearance <30mL/min

    Within 3 months of enrollment:
24. Significant gastrointestinal (GI) bleed
25. Myocardial infarction (MI), unstable angina, cardiac surgery or coronary intervention

    Within 6 months of enrollment:
26. Coronary artery bypass graft (CABG) procedure
27. Implant procedure performed for ICD, CRT leads or pacemaker
28. Documented stroke, CVA, TIA or suspected neurological event

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Atul Verma, MD, Principal Investigator — Medical Director, Heart Rhythm Program, Southlake Regional Health Centre; Andrea Natale, MD, Principal Investigator — Director, Electrophysiology, Texas Cardiac Arrhythmia Institute at St. David's Medical Center
Locations (28):
- United States (15):
  - Grandview Medical Center, Birmingham, Alabama
  - University Of Alabama, Birmingham, Alabama
  - Keck School Of Medicine, Los Angeles, California
  - Advent Health, Florida Hospital Orlando, Orlando, Florida
  - Iowa Heart Center, West Des Moines, Iowa
  - Kansas City Heart Rhythm Institute, Overland Park, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Jackson Heart Clinic, Jackson, Mississippi
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Medical Center, New York, New York
  - Trident Medical Center, Charleston, South Carolina
  - Medical University Of South Carolina, Charleston, South Carolina
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Houston Methodist Hospital, Houston, Texas
- Canada (3):
  - Southlake Regional Health Center, Newmarket, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec (IUCPQ), Québec, Quebec
- Czechia (3):
  - Institut Klinicke a Experimentalni Mediciny (IKEM), Prague, Czechia
  - Na Homolce, Prague, Prague
  - St Ann's University Hospital, Brno
- France (4):
  - Clinique du Tonkin, Villeurbanne, Lyon
  - CHRU Nancy, Nancy
  - Clinique Saint Pierre, Perpignan
  - Clinique Pasteur, Toulouse
- Leipzig Heart Institute GmbH, Leipzig, Germany
- Italy (2):
  - Centro Cardiologico Monzino, Milan, Milano
  - Ospedale dell'Angelo, Venezia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the study occurred from September 2018 to November 2023. The first subject was enrolled on September 19, 2018, and the last patient visit occurred on October 31, 2024.
Pre-assignment Details: Of the 376 subjects enrolled, 15 exited the study prior to undergoing ablation and were not included in the intent-to-treat (ITT) population. These subjects may have exited for various reasons including withdrawal of consent or clinical exclusion criteria discovered after enrollment. Baseline assessments were conducted prior to ablation to confirm eligibility and ensure protocol compliance.
Groups:
- Enrolled subjects: All enrolled subjects underwent catheter ablation using the DiamondTemp™ Ablation (DTA) system. A total of 376 subjects were enrolled.
Period: Overall Study
Arm/Group | Enrolled subjects
Started | 376
Intention-to-treat (ITT) (Of all enrolled subjects, 361 subjects underwent an ablation, forming the ITT cohort.) | 361
Modified intention-to-treat (MITT) (The mITT population (n=290) included subjects who met all eligibility criteria and were ablated.) | 290
Completed | 275
Not Completed | 101

BASELINE CHARACTERISTICS:
Groups:
- Modified Intention-to-treat (mITT) Cohort: All enrolled subjects underwent catheter ablation using the DiamondTemp™ Ablation (DTA) system. A total of 376 subjects were enrolled. Of these, 361 subjects underwent ablation and formed the intent-to-treat (ITT) population. Following ablation, subjects were followed for 12 months to assess safety and effectiveness outcomes. The mITT population (n=290) included subjects who met all eligibility criteria and were ablated.
  Subjects not meeting all eligibility criteria (n=71) were still followed as part of a secondary analysis. The follow-up protocol included scheduled assessments and monitoring at predetermined time points up to 12 months post-ablation.
  Exit reasons included voluntary withdrawal, death, or loss to follow-up.
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 290
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 216
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 231
  Unknown or Not Reported | 45
Race/Ethnicity, Customized [Number; unit: participants]
  African | 4
  Americas (Native North, South American, Canadian First) | 5
  Caucasian (European descent) | 228
  Unknown | 48
  Other | 7

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Events
Description: Participant count of a composite of safety events including: serious adverse events (SAEs), procedure and/or device-related significant pericardial effusion, severe or clinically symptomatic pulmonary vein stenosis and atrioesophageal fistula
Time Frame: Ablation through 6 months
Measure: Number; unit: participants
Groups:
- Modified Intention-to-treat (mITT) Cohort: Subjects who met all eligibility criteria and were ablated.
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 290
participants | 16

2. Primary Outcome: Primary Effectiveness
Description: The primary effectiveness endpoint is defined as freedom from documented AF, Atrial Flutter, (AFL) and Atrial Tachycardia (AT) episodes following the blanking period (3-month follow-up post-ablation procedure) through the end of the effectiveness evaluation period (12-month follow-up post-ablation procedure).
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 290
participants | 198

3. Secondary Outcome: Freedom From a Composite of Serious Adverse Events (SAEs)
Description: Freedom from a composite of SAEs occurring within 30-days post-index ablation procedure as adjudicated by an independent CEC for relatedness to the procedure or device.
Time Frame: Within 30-days post-index ablation
Measure: Number; unit: participants
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 290
participants | 273

4. Secondary Outcome: Freedom From Documented AF/AFL/AT Episodes
Description: Freedom from documented AF/AFL/AT episodes during the effectiveness evaluation period lasting ≥ 30 seconds in duration by ECG monitoring.
Time Frame: Within 3 months
Measure: Number; unit: participants
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 290
participants | 188

5. Secondary Outcome: Freedom From Documented AF/AFL/AT Episodes in the Absence of Class I and III Anti-arrhythmic Drug Therapy.
Description: Freedom from documented AF/AFL/AT episodes during the effectiveness evaluation period in the absence of class I and III anti-arrhythmic drug therapy.
Time Frame: Within 3 months
Measure: Number; unit: participants
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 290
participants | 126

6. Secondary Outcome: Acute Procedural Success
Description: Participant count of acute procedural success, defined as confirmation of electrical isolation of PVs via assessment of entrance block at least 20 minutes following the last ablation around the respective PV
Time Frame: Day of index ablation procedure
Measure: Number; unit: participants
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 290
participants | 289

7. Secondary Outcome: Single Procedure Success With Freedom From AF/AT/AFL
Description: Participant count of single procedure success defined as the rate of subjects treated with one single ablation procedure for the entire enrollment period and with freedom from documented symptomatic AF, AT and AFL* at 12 months.
Time Frame: 12 months after the index ablation procedure
Measure: Number; unit: participants
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 290
participants | 172

8. Secondary Outcome: Single Procedure Success With Freedom From All Primary Effectiveness Failures
Description: Participant count of single procedure success with freedom from all primary effectiveness failure criteria.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 290
participants | 155

9. Secondary Outcome: AFEQT Quality of Life, Baseline
Description: QOL using the AFEQT Questionnaire, baseline questionnaires.
  The scale is the AF Effect on Quality-of-Life (AFEQT) score. Higher scores are better. Minimum value: 0. Maximum value: 100.
Time Frame: Day of index ablation procedure
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 290
score on a scale | 61.6 [59.1 to 64.1]

10. Secondary Outcome: AFEQT Quality of Life, 6-month Follow-up
Description: QOL using the AFEQT Questionnaire, 6 month questionnaires.
  The scale is the AF Effect on Quality-of-Life (AFEQT) score. Higher scores are better. Minimum value: 0. Maximum value: 100.
Time Frame: 6 months after index ablation procedure
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 270
score on a scale | 85.6 [83.9 to 87.2]

11. Secondary Outcome: AFEQT Quality of Life, 12-month Follow up
Description: QOL using the AFEQT Questionnaire, 12-month questionnaires.
  The scale is the AF Effect on Quality-of-Life (AFEQT) score. Higher scores are better. Minimum value: 0. Maximum value: 100.
Time Frame: 12 months after index ablation procedure
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 274
score on a scale | 88.0 [86.1 to 89.8]

12. Secondary Outcome: Change in AFEQT Quality of Life From Baseline to 12-month
Description: Changes in QOL using the AFEQT Questionnaire between 12-month and baseline questionnaires.
  The scale is the AF Effect on Quality-of-Life (AFEQT) score. Higher scores are better. Minimum value: 0. Maximum value: 100.
Time Frame: Index ablation procedure through 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 274
score on a scale | 26.5 [23.8 to 29.2]

13. Secondary Outcome: National Institutes of Health Stroke Scale, Pre-discharge
Description: Neurological changes measured using the National Institutes of Health Stroke Scale (NIHSS)
  The NIHSS which is comprised of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score possible is 0.
Time Frame: Day of index ablation procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 286
Participants
  Improved -3 from baseline to pre-discharge | 0
  Stayed the same +0 from baseline to pre-discharge | 282
  Worsened +2 from baseline to pre-discharge | 1
  Worsened +1 from baseline to pre-discharge | 2
  Improved -2 from baseline to pre-discharge | 0
  Improved -1 from baseline to pre-discharge | 1

14. Secondary Outcome: National Institutes of Health Stroke Scale, One- Month Follow up
Description: as for outcome 13
Time Frame: One month after index ablation procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 198
Participants
  Improved -3 from baseline to 1-month follow-up | 0
  Stayed the same +0 from baseline to 1-month follow-up | 197
  Worsened +1 from baseline to 1-month follow-up | 0
  Improved -1 from baseline to 1-month follow-up | 1
  Worsened +2 from baseline to 1-month follow-up | 0
  Improved -2 from baseline to 1-month follow-up | 0

15. Secondary Outcome: National Institutes of Health Stroke Scale, 12-month Follow-up
Description: as for outcome 13
Time Frame: 12 months after the index ablation procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 237
Participants
  Improved -3 from baseline to 12-month follow-up | 1
  Worsened +2 from baseline to 12-month follow-up | 1
  Stayed the same +0 from baseline to 12-month follow-up | 228
  Improved -2 from baseline to 12-month follow-up | 0
  Improved -1 from baseline to 12-month follow-up | 4
  Worsened +1 from baseline to 12-month follow-up | 3

16. Other Pre Specified Outcome: Total Procedure Time (Minutes)
Description: Total procedure time (minutes), defined as time of investigational catheter insertion into the vasculature to time of last procedural ablation catheter removed.
Time Frame: Immediately after the index ablation procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 289
minutes | 104.0 (34.8)

17. Other Pre Specified Outcome: Total Treatment Device Time (Minutes)
Description: Total treatment device time (minutes), defined as time of delivery of first RF ablation with investigational catheter to removal of the investigational catheter.
Time Frame: Day of index ablation procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 289
minutes | 85.8 (31.8)

18. Other Pre Specified Outcome: Cumulative RF Time
Description: Mean cumulative RF Time (minutes).
Time Frame: Day of index ablation procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 288
minutes | 47.6 (34.8)

19. Other Pre Specified Outcome: Duration of RF Ablations (Seconds)
Description: Mean duration of RF ablations (seconds)
Time Frame: Day of index ablation procedure
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 279
seconds | 17.0 (22.2)

20. Other Pre Specified Outcome: Fluid Infused Through the Investigational Catheter (mL)
Description: Total fluid infused through the investigational catheter (mL)
Time Frame: Day of index ablation procedure
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 281
mL | 265.5 (121.9)

21. Other Pre Specified Outcome: Fluoroscopy Time (Minutes)
Description: Total fluoroscopy exposure time (minutes)
Time Frame: Day of index ablation procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 290
minutes | 13.6 (17.6)

22. Other Pre Specified Outcome: Incidence of Re-hospitalizations Due to Atrial Fibrillation Recurrence.
Description: Number of subjects who were re-hospitalized due to atrial fibrillation recurrence after blanking period.
Time Frame: Between the blanking period (3-month follow-up post-ablation procedure) through the end of the effectiveness evaluation period (12-month follow-up post-ablation procedure).
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Intention-to-treat (mITT) Cohort
Number analyzed (Participants) | 290
Participants
  0 Re-hospitalizations | 285
  1 Re-hospitalization | 5

ADVERSE EVENTS:
Time Frame: From index ablation procedure through 12 months of follow-up.
Groups:
- Intention-to-treat (ITT): There were 376 subjects enrolled in the study. Of these, 361 (96.0%) underwent an ablation, while 15 exited without undergoing ablation.
Arm/Group | Intention-to-treat (ITT)
All-Cause Mortality (participants affected / at risk) | 2/361
Serious Adverse Events (participants affected / at risk) | 78/361
Other Adverse Events (participants affected / at risk) | 22/361
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intention-to-treat (ITT) (N=361)
Anaemia (Blood and lymphatic system disorders) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2)
Angina unstable (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 11 (12)
Atrial flutter (Cardiac disorders) | 9 (9)
Atrial tachycardia (Cardiac disorders) | 6 (6)
Cardiac failure (Cardiac disorders) | 4 (4)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 3 (3)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 2 (2)
Right ventricular failure (Cardiac disorders) | 1 (1)
Sinus arrest (Cardiac disorders) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 2 (2)
Visual impairment (Eye disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 6 (6)
Implant site extravasation (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (3)
Graft infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Post procedural pneumonia (Infections and infestations) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 2 (2)
Streptococcal infection (Infections and infestations) | 1 (1)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1)
Post procedural stroke (Injury, poisoning and procedural complications) | 4 (4)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Migraine with aura (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Device pacing issue (Product Issues) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Haemorrhoid operation (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypertensive crisis (Vascular disorders) | 1 (1)
Hypertensive urgency (Vascular disorders) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intention-to-treat (ITT) (N=361)
Atrial Flutter (Cardiac disorders) | 22 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT03643224/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT03643224/SAP_001.pdf